CLINICAL TRIAL: NCT00558376
Title: Polyethylene Glycol Versus Sodium Phosphate for Colon Preparation After Failure of First Preparation for Colonoscopy - An Investigator Blinded Prospective Controlled Trial
Brief Title: Polyethylene Glycol Versus Sodium Phosphate for Colon Preparation After Failure of First Preparation for Colonoscopy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to FDA alert regarding Fleet phosphosoda
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Shomron BenHorin, Professor, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHEBA-07-4884-SBH-CTIL
Record Dates: First submitted 2007-11-13; First posted 2007-11-14 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Colonoscopy
Keywords: Colonoscopy
MeSH Terms: interventions — Polyethylene Glycols; polyethylene glycol 3350; sodium phosphate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Ingestion of 3L polyethylene Glycol
  Interventions: Drug: polyethylene glycol
- 2 (Active Comparator): Ingestion of 2 doses of sodium phosphate 45 cc
  Interventions: Drug: Sodium phosphate

INTERVENTIONS:
Drug: polyethylene glycol — Single time 3 liters PEG, 250 cc every 15 minutes the day before colonoscopy
  Other Names: Meroken New, Polyethylene glycol 3350, Taro, Israel
  Arms: 1
Drug: Sodium phosphate — Sodium phosphate 45cc, 2 doses 4 hours apart the day before colonoscopy
  Other Names: Sodium phosphate solution; Soffodex, Dexxon, Israel
  Arms: 2

SUMMARY:
The aim of the study is to compare the efficacy of Polyethylene glycol versus sodium phosphate as purgative for colon preparation to colonoscopy, after the failure of preparation with sodium phosphate for first colonoscopy. The hypothesis tested is whether there is advantage for substituting the purgative used, as compared to repeating the colonoscopy with the same purgative.Briefly, patients whose preparation was inadequate, will be allocated randomly to a group that will receive 3L Polyethylene glycol versus a group that will receive sodium phosphate(45ccX2). Both groups will be instructed to extend low-fiber diet to 5 days. Cleanliness of the colon at colonoscopy will be assessed blindly by an experienced endoscopist.

DETAILED DESCRIPTION:
The aim of the study is to compare the efficacy of Polyethylene glycol versus sodium phosphate as purgative for colon preparation to colonoscopy, after the failure of preparation with sodium phosphate for first colonoscopy. The hypothesis tested is whether there is advantage for substituting the purgative used, as compared to repeating the colonoscopy with the same purgative.Briefly, the study will be composed of patients whose preparation was judged to be inadequate in a first colonoscopy by an endoscopist independent of the current study. They will be allocated randomly to a group that will receive 3L Polyethylene glycol versus a group that will receive sodium phosphate(45ccX2). Both groups will be instructed to extend low-fiber diet to 5 days. Cleanliness of the colon at colonoscopy will be assessed blindly by an experienced endoscopist.

ELIGIBILITY:
Inclusion Criteria:

* Failed colonoscopy due to inadequate preparation
* Able to understand and sign an informed consent
* Preparation for frst colonoscopy consisted of sodium phosphate

Exclusion Criteria:

* Significant heart disease or CHF
* Chronic Renal Failure
* Allergy to any of the purgative ingredients
* Pregnancy
* Alcohol and/or drug abuse
* Vomiting or aspiration
* Suspected bowel obstruction

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Colon cleanliness at the second colonoscopy | within 24 hours of purgative ingestion, and within 30 minutes of colonoscopy

SECONDARY OUTCOMES:
Tolerability of purgative regimen | within 24 hours of purgative ingestion

CONTACTS AND LOCATIONS:
Overall Officials: Shomron Ben-Horin, MD, Principal Investigator — Sheba Medical Center; Benjamin Avidan, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba_Medical_Center, Tel Litwinsky, Israel